CLINICAL TRIAL: NCT03933202
Title: Cladribine Tablets: Observational Evaluation of Effectiveness and PROs in Suboptimally Controlled Patients Previously Taking Oral or Infusion DMDs for RMS (MASTER-2)
Brief Title: A Study of Suboptimally Controlled Participants Previously Taking Oral or Infusion DMDs for RMS (MASTER-2)
Status: Completed | Type: Observational
Sponsor: EMD Serono Research & Development Institute, Inc. (Industry)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Organization: EMD Serono (Industry)
Other Study IDs: MS700568_0079
Record Dates: First submitted 2019-04-29; First posted 2019-05-01 (Actual); Results first posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Cladribine Tablets; Observational; Mavenclad
MeSH Terms: conditions — Multiple Sclerosis | interventions — Cladribine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cladribine Tablets: No intervention will be administered as a part of this study. Participants who had decided prior to enrollment to transition from any oral or infusion DMD to treatment with cladribine tablets under routine clinical care and who meet all eligibility criteria will receive an initial treatment course with cladribine tablets in Year 1 and are planned to receive a second course in Year 2, as per the approved United States Prescribing Information (USPI). Data sources for this study will include data extracts from participants' medical records performed by site personnel as well as questionnaires directly filled out by participants.
  Interventions: Drug: Cladribine Tablets

INTERVENTIONS:
Drug: Cladribine Tablets — No intervention will be administered as a part of this study. Participants will receive cladribine tablets as per investigator discretion and as per United States approved label: 3.5 milligram/kilogram (mg/kg) body weight over 2 years, administered as 1 treatment course of 1.75 mg/kg per year.

SUMMARY:
To evaluate the effectiveness, safety and Patient-Reported Outcomes (PROs) of cladribine tablets in participants with RMS including relapsing-remitting multiple sclerosis (RRMS) and active secondary progressive multiple sclerosis (aSPMS), who transition to cladribine tablets after suboptimal response to any oral or infusion Disease-Modifying Drugs (DMDs) approved in the United States (US) for RMS in a real-world-setting.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Have diagnosis of RMS, including RRMS and aSPMS, and satisfy the approved indication for cladribine tablets as per United States Prescribing Information (USPI)
* Have time since diagnosis of RMS of at least 12 months
* In the opinion of the investigator, experienced suboptimal response (lack of effectiveness, intolerability, poor adherence) to oral or infusion DMD treatment other than cladribine tablets
* Had received their last previous oral DMD for at least 1 month or at least 1 dose of their last previous infusion DMD
* Have decided to initiate treatment with cladribine tablets during routine clinical care
* Meet criteria as per the approved USPI
* Have access to a valid e-mail address

Exclusion Criteria:

* Have been previously treated with cladribine in any dosing form (intravenous, subcutaneous, or oral)
* Transitioning from previous oral DMD solely for administrative reasons such as relocation
* Have comorbid conditions that preclude participation
* Have any clinical condition or medical history noted as contraindication on USPI
* Are currently participating in an interventional clinical trial
* Pregnant or breastfeeding women, women who plan to become pregnant or men whose partner plans to become pregnant during study the cladribine treatment period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with relapsing form of Multiple Sclerosis (RMS) including active secondary progressive multiple sclerosis (aSPMS).
Sampling Method: Non-Probability Sample
Enrollment: 291 (Actual)
Dates: Start 2019-07-22 (Actual); Primary Completion 2024-11-11 (Actual); Study Completion 2024-11-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — EMD Serono Inc., the biopharmaceutical division of Merck KGaA, Darmstadt, Germany
Locations (66):
- United States (66):
  - North Central Neurology Associates, P.C., Cullman, Alabama
  - University of South Alabama, Mobile, Alabama
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Fullerton Neurology and Headache Center, Fullerton, California
  - Regina Berkovich MD PhD INC, West Hollywood, California
  - Colorado Springs Neurological Associates, PC - Neurology, Colorado Springs, Colorado
  - HCA Research Institute, Englewood, Colorado
  - Advanced Neurosciences Research, LLC, Fort Collins, Colorado
  - Associated Neurologists of Southern Connecticut, PC, Fairfield, Connecticut
  - Yale University, Fairfield, Connecticut
  - Neurology Associates, P. A., Maitland, Florida
  - University of Miami, Miami, Florida
  - Orlando Health Multiple Sclerosis Comprehensive Care Center - Downtown Orlando, Orlando, Florida
  - Suncoast Neuroscience and Associates, Inc., St. Petersburg, Florida
  - Axiom Clinical Research of Florida, Tampa, Florida
  - University of South Florida, Tampa, Florida
  - Northwest Neurology Ltd, Rolling Meadows, Illinois
  - Prairie Education & Research, Springfield, Illinois
  - Fort Wayne Neurological Center, Fort Wayne, Indiana
  - College Park Family Care Center, Overland Park, Kansas
  - Baptist Health Lexington, Lexington, Kentucky
  - Northern Light Comprehensive Multiple Sclerosis Care Center, Bangor, Maine
  - Neurological Clinical Research Institute, Boston, Massachusetts
  - Neuro Institute of New England P.C., Foxborough, Massachusetts
  - The Elliot Lewis Center for Multiple Sclerosis Care, Wellesley, Massachusetts
  - UMASS - Neurology, Worcester, Massachusetts
  - Wayne State University (WSU) - Multiple Sclerosis Treatment and Clinical Research Center (MS Center) - Department of Neurology, Detroit, Michigan
  - Detroit Clinical Research Center, PC, Farmington Hills, Michigan
  - Memorial Healthcare, Owosso, Michigan
  - Minneapolis Clinic of Neurology - Neurology, Golden Valley, Minnesota
  - Neurology Center of Las Vegas, Las Vegas, Nevada
  - DENT Neurologic Institute, Amherst, New York
  - NYU Langone Brooklyn - Brooklyn, Brooklyn, New York
  - The Trustee of Columbia University in the City of New York, New York, New York
  - The Charlotte-Mecklenburg Hospital Authority - Carolinas Healthcare System, Charlotte, North Carolina
  - Guilford Neurologic Associates, Greensboro, North Carolina
  - Raleigh Neurology Associates, Raleigh, North Carolina
  - Insight Neuroscience LLC, Bellevue, Ohio
  - Riverhills Neuroscience, Cincinnati, Ohio
  - The Boster Center for Multiple Scelosis, Columbus, Ohio
  - Dayton Center for Neurological Disorders, Dayton, Ohio
  - University of Toledo - PARENT, Toledo, Ohio
  - Providence Neurological Specialties, Portland, Oregon
  - Wills Eye Institute - Ocular Oncology Service - Wills Eye Institute, Philadelphia, Pennsylvania
  - Premier Neurology Research, P.C., Greer, South Carolina
  - Neurology, PC, Knoxville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Northwest Houston Neurology, Cypress, Texas
  - Baylor College of Medicine IRB, Houston, Texas
  - DHR Health Neurology Institute Neuroimmunology and Multiple Sclerosis, McAllen, Texas
  - Central Texas Neurology Consultants, Round Rock, Texas
  - Neurology Center of San Antonio, San Antonio, Texas
  - Integrated Neurology Services - Dr. Simon Fishman's Office, Alexandria, Virginia
  - Blacksburg Neurology, PC, Christiansburg, Virginia
  - Meridian Clinical Research (Neurology), Norfolk, Virginia
  - Neurological Associates, Richmond, Virginia
  - VCU Medical Center - Pediatric Neurology, Richmond, Virginia
  - Massey Cancer Center - VCU Medical Center, Richmond, Virginia
  - Multiple Sclerosis Center of Greater Washington, Vienna, Virginia
  - Sentara Ambulatory Care Center, Virginia Beach, Virginia
  - MS Center of Evergreen, Kirkland, Washington
  - MultiCare Health System Institute for Research and Innovation - MultiCare Health System Institute for Research and, Spokane, Washington
  - MultiCare Health System Institute for Research and Innovation - MultiCare Health System Institute for Research, Tacoma, Washington
  - Ascension St. Francis Center for Neurological Disorders, S.C., Milwaukee, Wisconsin
  - The Medical College of Wisconsin - Endocrinology, Milwaukee, Wisconsin
  - Neuroscience Group of Northeast Wisconsin - DUPLICATE, Neenah, Wisconsin

REFERENCES:
- [Derived] Miravalle AA, Katz J, Robertson D, Hayward B, Harlow DE, Lebson LA, Sloane JA, Bass AD, Fox EJ. CLICK-MS and MASTER-2 Phase IV trial design: cladribine tablets in suboptimally controlled relapsing multiple sclerosis. Neurodegener Dis Manag. 2021 Apr;11(2):99-111. doi: 10.2217/nmt-2020-0059. Epub 2021 Feb 1. PMID 33517769
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=MS700568_0079
- See also: US Medical Information website, Medical Resources — https://medical.emdserono.com/en_US/home.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Cladribine Tablets: Switch From Oral: Participants who had decided prior to enrollment to transition from any oral Disease-Modifying Drug (DMD) to treatment with cladribine tablets under routine clinical care and who met all eligibility criteria received an initial treatment course with cladribine tablets in Year 1 and a second course in Year 2, as per the approved United States Prescribing Information (USPI). No intervention was administered as a part of this study and all data was prospectively collected during this study.
- Cladribine Tablets: Switch From Infusion: Participants who had decided prior to enrollment to transition from any infusion DMD to treatment with cladribine tablets under routine clinical care and who met all eligibility criteria received an initial treatment course with cladribine tablets in Year 1 and a second course in Year 2, as per the approved United States Prescribing Information (USPI). No intervention was administered as a part of this study and all data was prospectively collected during this study.
Period: Overall Study
Arm/Group | Cladribine Tablets: Switch From Oral | Cladribine Tablets: Switch From Infusion
Started | 163 | 120
Participants Who Received at Least 1 Dose of Cladribine Tablets | 103 | 85
Switch From Ocrelizumab (Participants who switched from infusion DMD (ocrelizumab) to CladT) | 0 | 53
Completed | 116 | 92
Not Completed | 47 | 28
Not completed — Participant withdrawn by Principal Investigator | 1 | 0
Not completed — Participant transferred care | 1 | 0
Not completed — Site research department closing | 1 | 0
Not completed — Site closed prematurely due to unexpected circumstances | 0 | 1
Not completed — Participant discontinuation due to Sponsor decision to close study | 0 | 2
Not completed — Participant changed primary neurology provider | 1 | 0
Not completed — Participant could not be entered as a follow-up | 0 | 1
Not completed — Participant non-compliant, therefore, has been discontinued | 1 | 0
Not completed — Participant delayed year 2 due to subject fear of COVID-19 | 1 | 0
Not completed — Missed visit | 0 | 1
Not completed — Investigator decision | 4 | 0
Not completed — Discontinuation due to safety extension removal by Sponsor | 0 | 1
Not completed — Withdrawal by Subject | 10 | 8
Not completed — Death | 2 | 0
Not completed — Progressive disease | 0 | 3
Not completed — Protocol non-compliance | 6 | 3
Not completed — Lost to Follow-up | 16 | 8
Not completed — Adverse Event | 3 | 0

BASELINE CHARACTERISTICS:
Population: FAS included all participants enrolled in the study who received at least 1 dose of cladribine tablets.
Groups:
- Cladribine Tablets: Switch From Oral: Participants who had decided prior to enrollment to transition from any oral DMD to treatment with cladribine tablets under routine clinical care and who met all eligibility criteria received an initial treatment course with cladribine tablets in Year 1 and a second course in Year 2, as per the approved United States Prescribing Information (USPI). No intervention was administered as a part of this study and all data was prospectively collected during this study.
- Total: Total of all reporting groups
Arm/Group | Cladribine Tablets: Switch From Oral | Cladribine Tablets: Switch From Infusion | Total
Number analyzed (Participants) | 103 | 85 | 188
Age, Continuous [Mean (Standard Deviation); unit: years] | 50 (10.8) | 48 (12.5) | 49 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 84 | 58 | 142
  Male | 19 | 27 | 46
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 3 | 8
  Not Hispanic or Latino | 93 | 74 | 167
  Unknown or Not Reported | 5 | 8 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 13 | 6 | 19
  White | 85 | 68 | 153
  More than one race | 0 | 4 | 4
  Unknown or Not Reported | 4 | 5 | 9

OUTCOME MEASURES:

1. Secondary Outcome: Change From Baseline in 14-Item Treatment Satisfaction Questionnaire for Medication (TSQM-14) Score at Month 6, 12 and 24
Description: The TSQM-14 was a participant-rated scale used to assess subjective satisfaction with medication. The TSQM has 14 questions that assesses participants' global satisfaction level with their treatment in 4 domains: side effects (There are 5 questions in the side effects domain, however one of them is a Yes/No question and there are 4 sub-components, hence a maximum score of 20), effectiveness (3 questions), global satisfaction (3 questions), and convenience (3 questions). All questions are scored from 1 (least satisfied) to 5 or 7 (most satisfied). The total score is summed for each domain to obtain: side effects (1-20), effectiveness (1-21), global satisfaction (1-17), and convenience (1-21), using transformed scores between 0 and 100. Lower total scores in each domain indicate dissatisfaction with the study medication and higher total scores indicate satisfaction.
Time Frame: Baseline (Month 0), Month 6, 12 and 24
Population: The FAS included all participants enrolled in the study who received at least 1 dose of cladribine tablets. "Overall number of participants analyzed" refers to those evaluable for the outcome measure, while "number analyzed" refers to those evaluable at specific timepoints.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cladribine Tablets: Switch From Oral | Cladribine Tablets: Switch From Infusion
Number analyzed (Participants) | 46 | 29
units on a scale
  Global Satisfaction: Month 6: number analyzed (Participants) | 17 | 7
  Global Satisfaction: Month 6 | 18.5 (30.42) | 22.2 (15.14)
  Global Satisfaction: Month 12: number analyzed (Participants) | 18 | 3
  Global Satisfaction: Month 12 | 11.1 (25.95) | 19.0 (21.82)
  Global Satisfaction: Month 24: number analyzed (Participants) | 4 | 1
  Global Satisfaction: Month 24 | 16.1 (24.31) | -28.6 (NA) — Standard deviation could not be calculated due to high missingness and low response rate.
  Effectiveness: Month 6: number analyzed (Participants) | 17 | 6
  Effectiveness: Month 6 | 10.5 (29.13) | 22.2 (21.08)
  Effectiveness: Month 12: number analyzed (Participants) | 18 | 3
  Effectiveness: Month 12 | 3.9 (24.09) | 24.1 (30.60)
  Effectiveness: Month 24: number analyzed (Participants) | 4 | 1
  Effectiveness: Month 24 | 2.8 (21.52) | 16.7 (NA) — Standard deviation could not be calculated due to high missingness and low response rate.
  Side Effects: Month 6: number analyzed (Participants) | 17 | 7
  Side Effects: Month 6 | 11.4 (40.28) | 7.1 (16.31)
  Side Effects: Month 12: number analyzed (Participants) | 18 | 3
  Side Effects: Month 12 | 6.3 (24.63) | 2.1 (40.67)
  Side Effects: Month 24: number analyzed (Participants) | 4 | 0
  Side Effects: Month 24 | 10.9 (12.88) |
  Convenience: Month 6: number analyzed (Participants) | 17 | 7
  Convenience: Month 6 | 15.4 (27.25) | 24.6 (14.29)
  Convenience: Month 12: number analyzed (Participants) | 18 | 3
  Convenience: Month 12 | 7.7 (29.90) | 18.5 (28.51)
  Convenience: Month 24: number analyzed (Participants) | 4 | 1
  Convenience: Month 24 | 1.4 (53.74) | 44.4 (NA) — Standard deviation could not be calculated due to high missingness and low response rate.

2. Secondary Outcome: Change From Baseline in 36-Item Short Form Health Survey (SF-36) Domain Score at Month 6, 12 and 24
Description: The SF-36 Health Survey is a validated, self-administered questionnaire designed to assess general health status across eight domains: physical functioning, role limitations due to physical health, bodily pain, general health perceptions, vitality, social functioning, role limitations due to emotional problems, and mental health. It includes one item evaluating perceived change in health over the past year and generates two summary scores-the Physical Component Summary (PCS) and Mental Component Summary (MCS)-derived using factor analytic methods. Each domain and summary score is scaled from 0 to 100, with higher scores indicating better health status.
Time Frame: Baseline (Month 0), Month 6, 12 and 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cladribine Tablets: Switch From Oral | Cladribine Tablets: Switch From Infusion
Number analyzed (Participants) | 61 | 46
units on a scale
  PCS: Baseline | 44.2 (11.17) | 38.1 (10.76)
  PCS: Month 6: number analyzed (Participants) | 22 | 12
  PCS: Month 6 | 0.4 (5.43) | 2.2 (6.75)
  PCS: Month 12: number analyzed (Participants) | 24 | 6
  PCS: Month 12 | 0.2 (6.44) | -1.9 (5.54)
  PCS: Month 24: number analyzed (Participants) | 9 | 3
  PCS: Month 24 | 1.0 (6.06) | -2.0 (6.94)
  MCS: Baseline | 48.2 (9.35) | 46.4 (12.01)
  MCS: Month 6: number analyzed (Participants) | 22 | 12
  MCS: Month 6 | 2.3 (8.63) | -1.6 (6.45)
  MCS: Month 12: number analyzed (Participants) | 24 | 6
  MCS: Month 12 | 0.8 (7.98) | -2.9 (4.70)
  MCS: Month 24: number analyzed (Participants) | 9 | 3
  MCS: Month 24 | -0.6 (8.77) | 2.8 (10.42)

3. Secondary Outcome: Change From Baseline in Modified Fatigue Impact Scale - 5-item Version (MFIS-5) Total Score at Month 6, 12 and 24
Description: The MFIS-5 is a shortened version of the Fatigue Impact Scale consisting of 5 items that assess the impact of fatigue on physical, cognitive, and psychosocial functioning. Each item is rated on a 5-point Likert scale: 0 (Never), 1 (Rarely), 2 (Sometimes), 3 (Often), and 4 (Almost always). The total score ranges from 0 to 20, with higher scores indicating a greater impact of fatigue. Items include: reduced alertness, limitations in activities away from home, difficulty sustaining physical effort, reduced ability to complete tasks requiring physical effort, and trouble concentrating.
Time Frame: Baseline (Month 0), Month 6, 12 and 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cladribine Tablets: Switch From Oral | Cladribine Tablets: Switch From Infusion
Number analyzed (Participants) | 54 | 37
units on a scale
  Baseline | 9.0 (5.14) | 10.5 (5.22)
  Month 6: number analyzed (Participants) | 21 | 10
  Month 6 | 0.0 (2.43) | -0.8 (3.52)
  Month 12: number analyzed (Participants) | 21 | 4
  Month 12 | -0.3 (2.87) | 1.5 (1.00)
  Month 24: number analyzed (Participants) | 7 | 2
  Month 24 | 0.9 (3.29) | 2.0 (1.41)

4. Secondary Outcome: Change From Baseline in 7-Item Beck-Depression Inventory-Fast Screen (BDI-FS) Total Score at Month 6, 12 and 24
Description: The 7-item Beck Depression Inventory-Fast Screen (BDI-FS) is a self-report tool used to assess the severity of depressive symptoms. It includes seven items: Sadness, Pessimism, Past Failure, Loss of Pleasure, Self-Dislike, Self-Criticalness, and Suicidal Thoughts. Each item is rated on a 4-point scale from 0 to 3, with higher scores indicating greater symptom severity. The total score ranges from 0 to 21 and is calculated by summing the highest-rated response for each item.
Time Frame: Baseline (Month 0), Month 6, 12 and 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cladribine Tablets: Switch From Oral | Cladribine Tablets: Switch From Infusion
Number analyzed (Participants) | 54 | 38
units on a scale
  Baseline | 1.8 (2.08) | 3.5 (3.55)
  Month 6: number analyzed (Participants) | 22 | 10
  Month 6 | 0.5 (1.54) | 1.0 (1.70)
  Month 12: number analyzed (Participants) | 22 | 4
  Month 12 | 0.2 (1.77) | 1.0 (2.16)
  Month 24: number analyzed (Participants) | 9 | 3
  Month 24 | 0.8 (1.48) | 0.3 (2.52)

5. Secondary Outcome: Change From Baseline in Percentage of Work Time Missed Assessed by 6-Item Work Productivity Activity Impairment - Multiple Sclerosis (WPAI-MS) Score at Month 6, 12 and 24
Description: The WPAI-MS questionnaire is a 6-item validated instrument to measure impairments in work and activities. The WPAI-MS included 6 questions: 1 (if currently employed); 2 (hours missed due to disease); 3 (hours missed other reasons); 4 (hours actually worked); 5 (degree disease affected productivity while working); 6 (degree disease affected regular activities). WPAI-MS generated four component scores: percentage of work time missed (absenteeism); percentage of impairment while working (presentisms); percentage of overall work impairment (absenteeism and presentisms combined); and percentage of activity impairment. Scores for WPAI range from 0% to 100%, where 0 % indicates no impairment and 100% is total loss of work productivity/activity. Change from baseline in percentage of work time missed (absenteeism) was reported.
Time Frame: Baseline (Month 0), Month 6, 12 and 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of work time missed
Arm/Group | Cladribine Tablets: Switch From Oral | Cladribine Tablets: Switch From Infusion
Number analyzed (Participants) | 16 | 6
percentage of work time missed
  Change at Month 6: number analyzed (Participants) | 14 | 6
  Change at Month 6 | 0.0 (39.22) | -8.7 (17.76)
  Change at Month 12: number analyzed (Participants) | 16 | 3
  Change at Month 12 | -7.7 (25.46) | 30.8 (60.08)
  Change at Month 24: number analyzed (Participants) | 7 | 1
  Change at Month 24 | 0.00 (0.00) | -100.0 (NA) — Standard deviation could not be calculated due to high missingness and low response rate.

6. Secondary Outcome: Change From Baseline in Percentage of Impairment While Working Assessed by 6-Item Work Productivity Activity Impairment - Multiple Sclerosis (WPAI-MS) Score at Month 6, 12 and 24
Description: The WPAI-MS questionnaire is a 6-item validated instrument to measure impairments in work and activities. The WPAI-MS included 6 questions: 1 (if currently employed); 2 (hours missed due to disease); 3 (hours missed other reasons); 4 (hours actually worked); 5 (degree disease affected productivity while working); 6 (degree disease affected regular activities). WPAI-MS generated four component scores: percentage of work time missed (absenteeism); percentage of impairment while working (presentisms); percentage of overall work impairment (absenteeism and presentisms combined); and percentage of activity impairment. Scores for WPAI range from 0% to 100%, where 0 % indicates no impairment and 100% is total loss of work productivity/activity. Change from baseline in percentage of impairment while working (presentisms) was reported.
Time Frame: Baseline (Month 0), Month 6, 12 and 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of impairment while working
Arm/Group | Cladribine Tablets: Switch From Oral | Cladribine Tablets: Switch From Infusion
Number analyzed (Participants) | 10 | 1
percentage of impairment while working
  Change at Month 6: number analyzed (Participants) | 9 | 1
  Change at Month 6 | -10.0 (16.58) | -10.0 (NA) — Standard deviation could not be calculated due to high missingness and low response rate.
  Change at Month 12 | -10.0 (34.32) | 0.0 (NA) — Standard deviation could not be calculated due to high missingness and low response rate.
  Change at Month 24: number analyzed (Participants) | 6 | 0
  Change at Month 24 | -1.7 (18.35) |

7. Secondary Outcome: Change From Baseline in Percentage of Overall Work Impairment Assessed by 6-Item Work Productivity Activity Impairment - Multiple Sclerosis (WPAI-MS) Score at Month 6, 12 and 24
Description: The WPAI-MS questionnaire is a 6-item validated instrument to measure impairments in work and activities. The WPAI-MS included 6 questions: 1 (if currently employed); 2 (hours missed due to disease); 3 (hours missed other reasons); 4 (hours actually worked); 5 (degree disease affected productivity while working); 6 (degree disease affected regular activities). WPAI-MS generated four component scores: percentage of work time missed (absenteeism); percentage of impairment while working (presentisms); percentage of overall work impairment (absenteeism and presentisms combined); and percentage of activity impairment. Scores for WPAI range from 0% to 100%, where 0 % indicates no impairment and 100% is total loss of work productivity/activity. Change from baseline in total percentage of work impairment (absenteeism and presentisms) were reported.
Time Frame: Baseline (Month 0), Month 6, 12 and 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of overall work impairment
Arm/Group | Cladribine Tablets: Switch From Oral | Cladribine Tablets: Switch From Infusion
Number analyzed (Participants) | 10 | 1
percentage of overall work impairment
  Change at Month 6: number analyzed (Participants) | 9 | 1
  Change at Month 6 | -10.0 (16.58) | -10.0 (NA) — Standard deviation could not be calculated due to high missingness and low response rate.
  Change at Month 12 | -9.8 (34.40) | 0.0 (NA) — Standard deviation could not be calculated due to high missingness and low response rate.
  Change at Month 24: number analyzed (Participants) | 6 | 0
  Change at Month 24 | -1.7 (18.35) |

8. Secondary Outcome: Change From Baseline in Percentage of Activity Impairment Assessed by 6-Item Work Productivity Activity Impairment- Multiple Sclerosis (WPAI-MS) Score at Month 6, 12 and 24
Description: The WPAI-MS questionnaire is a 6-item validated instrument to measure impairments in work and activities. The WPAI-MS included 6 questions: 1 (if currently employed); 2 (hours missed due to disease); 3 (hours missed other reasons); 4 (hours actually worked); 5 (degree disease affected productivity while working); 6 (degree disease affected regular activities). WPAI-MS generated four component scores: percentage of work time missed (absenteeism); percentage of impairment while working (presentisms); percentage of overall work impairment (absenteeism and presentisms combined); and percentage of activity impairment. Scores for WPAI range from 0% to 100%, where 0 % indicates no impairment and 100% is total loss of work productivity/activity. Change from baseline in percentage of activity impairment was reported.
Time Frame: Baseline (Month 0), Month 6, 12 and 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of activity impairment
Arm/Group | Cladribine Tablets: Switch From Oral | Cladribine Tablets: Switch From Infusion
Number analyzed (Participants) | 20 | 9
percentage of activity impairment
  Change at Month 6 | 3.5 (27.58) | -8.9 (18.33)
  Change at Month 12: number analyzed (Participants) | 18 | 4
  Change at Month 12 | -12.2 (23.40) | 10.0 (14.14)
  Change at Month 24: number analyzed (Participants) | 8 | 2
  Change at Month 24 | 0.0 (18.52) | -10.0 (14.14)

9. Secondary Outcome: Change From Baseline in Patient Determined Disease Steps (PDDS) Scale Total Score at Month 6, 12 and 24
Description: The PDDS is a patient-reported scale to assess the disability status in participants with MS, and it focuses mainly on how participants walk. Scores on the PDDS range from 0 (normal) to 8 (bedridden): 0 (Normal), 1 (Mild Disability), 2 (Moderate Disability), 3 (Gait Disability), 4 (Early Cane), 5 (Late Cane), 6 (Bilateral Support), 7 (Wheelchair/Scooter), and 8 (Bedridden). A higher score represents higher level of disability.
Time Frame: Baseline (Month 0), Month 6, 12 and 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cladribine Tablets: Switch From Oral | Cladribine Tablets: Switch From Infusion
Number analyzed (Participants) | 61 | 45
units on a scale
  Baseline | 2.1 (2.7) | 3.4 (2.47)
  Month 6: number analyzed (Participants) | 40 | 21
  Month 6 | -0.1 (1.01) | -0.4 (0.67)
  Month 12: number analyzed (Participants) | 34 | 19
  Month 12 | 0.0 (0.87) | -0.1 (0.81)
  Month 24: number analyzed (Participants) | 21 | 11
  Month 24 | -0.2 (1.04) | 0.0 (1.10)

10. Secondary Outcome: Number of Participants With Adherence to Treatment as Assessed by Modified Versions of the Multiple Sclerosis Treatment Adherence Questionnaire (MS-TAQ)
Description: 7 Treatment adherence questions, based on MS-TAQ, were developed to determine level of adherence as well as identify barriers to adherence for MS participants taking DMDs. 1.What treatment week of cladribine (Clad.) tablets (tab.) did you most recently complete? 2.How many Clad. tab. were you supposed to take during this treatment week? 3.Did you miss/forget to take any Clad. tab. during this treatment week? 4. How many Clad. tab. did you miss/ forget to take? 5.How important were following factors in missing/forgetting to take a dose? (scale from 0-3, where, 0=Not important at all and 3=Extremely important). 6.Overall, how hard/easy do you feel it is to take Clad. tab. as recommended by your physician during your treatment week? (scale from 1- 5, where 1=Extremely easy and 5=Extremely hard). 7.How satisfied are you with how things have been with your Clad. tab. treatment during your treatment week? (scale from 1-5, where 1=Not satisfied at all and 5=Completely satisfied).
Time Frame: Month 1, 2, 13 and 14
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cladribine Tablets: Switch From Oral | Cladribine Tablets: Switch From Infusion
Number analyzed (Participants) | 74 | 53
Participants
  Month 1: number analyzed (Participants) | 73 | 50
  Month 1 | 71 | 50
  Month 2 | 72 | 53
  Month 13: number analyzed (Participants) | 33 | 23
  Month 13 | 32 | 22
  Month 14: number analyzed (Participants) | 20 | 11
  Month 14 | 20 | 11

11. Secondary Outcome: Number of Participants Who Experienced Relapse
Description: A relapse was defined as per routine clinical practice as determined by the investigator. As a guide, relapse may be defined as exacerbation of symptoms that occur over a minimum of 24 hours and separated from a previous attack by at least 30 days, in the absence of fever or infection.
Time Frame: Over the 12-month and 24-month period
Population: The FAS included all participants enrolled in the study who received at least 1 dose of cladribine tablets.
Measure: Count of Participants; unit: Participants
Arm/Group | Cladribine Tablets: Switch From Oral | Cladribine Tablets: Switch From Infusion
Number analyzed (Participants) | 103 | 85
Participants
  Over the 12-month period | 4 | 4
  Over the 24-month period | 6 | 4

12. Secondary Outcome: Percentage of Participants With Relapse Associated With Hospitalization
Description: A relapse was defined according to routine clinical practice as determined by the investigator. A relapse will be associated with hospitalization if the participants will be hospitalized for the relapse. As a guide, relapse was considered an exacerbation of symptoms that occurred over a minimum of 24 hours and was separated from a previous attack by at least 30 days, in the absence of fever or infection. The percentage of participants who experienced a relapse associated with hospitalization was reported.
Time Frame: Over the 12-month period, 13th to 24th month and over the 24 month period.
Population: The FAS included all participants enrolled in the study who received at least 1 dose of cladribine tablets.
Measure: Number; unit: percentage of participants
Arm/Group | Cladribine Tablets: Switch From Oral | Cladribine Tablets: Switch From Infusion
Number analyzed (Participants) | 103 | 85
percentage of participants
  Over the 12-month period | 1.0 | 0.0
  13th to 24th month period | 0 | 0.0
  Over the 24-month period | 1.0 | 0.0

13. Secondary Outcome: Annualized Relapse Rate (ARR) Associated With Hospitalization at Months 12 and 24
Description: The qualifying relapse is the occurrence of new or worsening neurological symptoms attributable to Multiple Sclerosis (MS) (for more than [>] 24 hours, no fever, infection, injury, adverse events (AEs), and preceded by a stable or improving neurological state for more than or equal to [>=] 30 days).ARR was calculated as the total number of reported relapses in the 24 months after treatment divided by the days on study corresponding to relapse information and multiplied by 365.25. ARR associated with hospitalization at Months 12 and 24 were reported. A relapse was associated with hospitalization if the participant will be hospitalized for the relapse.
Time Frame: Month 12 and Month 24
Population: The FAS included all participants enrolled in the study who received at least 1 dose of cladribine tablets. Here, "overall Number of participants analyzed" signifies those participants who were evaluable for this outcome measure and "number analyzed" signifies those participants who were evaluable at each specified timepoints.
Measure: Mean (Standard Deviation); unit: relapses per year
Arm/Group | Cladribine Tablets: Switch From Oral | Cladribine Tablets: Switch From Infusion
Number analyzed (Participants) | 76 | 72
relapses per year
  Month 12 | 0.01 (0.114) | 0.00 (0.00)
  Month 24 | 0.01 (0.057) | 0.00 (0.00)

14. Secondary Outcome: Percentage of Participants With Relapse Associated With Glucocorticoid Use
Description: A relapse was defined according to routine clinical practice as determined by the investigator. As a guide, relapse was considered an exacerbation of symptoms that occurred over a minimum of 24 hours and was separated from a previous attack by at least 30 days, in the absence of fever or infection. The percentage of participants with relapse associated with glucocorticoid use over the 12-month period, 13th to 24th month and over the 24-month period of treatment with cladribine tablets was reported.
Time Frame: Over the 12-month period, 13th to 24th month and over the 24 month period.
Population: as for outcome 13
Measure: Number; unit: percentage of participants
Arm/Group | Cladribine Tablets: Switch From Oral | Cladribine Tablets: Switch From Infusion
Number analyzed (Participants) | 103 | 85
percentage of participants
  Over the 12-month period | 1.0 | 3.5
  13th to 24th month period | 1.0 | 0.0
  Over the 24-month period | 1.9 | 2.4

15. Secondary Outcome: Annualized Relapse Rate (ARR) Associated With Glucocorticoid Use at Months 12 and 24
Description: The qualifying relapse is the occurrence of new or worsening neurological symptoms attributable to Multiple Sclerosis (MS) (for more than [>] 24 hours, no fever, infection, injury, adverse events (AEs), and preceded by a stable or improving neurological state for more than or equal to [>=] 30 days). ARR was calculated as the total number of reported relapses in the 24 months after treatment divided by the days on study corresponding to relapse information and multiplied by 365.25. ARR associated with glucocorticoid use at Months 12 and 24 were reported. A relapse will be associated with glucocorticoid use if steroid treatment will be required for the relapse.
Time Frame: Months 12 and 24
Population: The FAS included all participants enrolled in the study who received at least 1 dose of cladribine tablets.
Measure: Mean (Standard Deviation); unit: relapses per year
Arm/Group | Cladribine Tablets: Switch From Oral | Cladribine Tablets: Switch From Infusion
Number analyzed (Participants) | 76 | 72
relapses per year
  Month 12 | 0.01 (0.114) | 0.04 (0.201)
  Month 24 | 0.02 (0.093) | 0.03 (0.142)

16. Secondary Outcome: Number of Previous Disease-Modifying Drugs (DMD) Received for Multiple Sclerosis (MS) at Baseline
Description: Number of previous DMD received by participants with MS were reported.
Time Frame: At Baseline (Month 0)
Population: The FAS included all participants enrolled in the study who received at least 1 dose of cladribine tablets.
Measure: Mean (Standard Deviation); unit: number of DMDs received
Arm/Group | Cladribine Tablets: Switch From Oral | Cladribine Tablets: Switch From Infusion
Number analyzed (Participants) | 103 | 85
number of DMDs received | 3.0 (1.66) | 3.4 (1.82)

17. Secondary Outcome: Percentage of Participants Who Discontinued Cladribine Tablets
Description: Percentage of participants who discontinued cladribine tablets were reported.
Time Frame: Baseline (Month 0) up to 24 Months
Population: The FAS included all participants enrolled in the study who received at least 1 dose of cladribine tablets.
Measure: Number; unit: percentage of participants
Arm/Group | Cladribine Tablets: Switch From Oral | Cladribine Tablets: Switch From Infusion
Number analyzed (Participants) | 103 | 85
percentage of participants | 41.7 | 22.4

18. Secondary Outcome: Number of Participants With Reason for Discontinuation of Cladribine Tablets
Description: Number of participants who discontinued cladribine tablets in each category of reason for discontinuation were reported.
Time Frame: Baseline (Month 0) up to 24 Months
Population: The FAS included all participants enrolled in the study who received at least 1 dose of cladribine tablets.
Measure: Count of Participants; unit: Participants
Arm/Group | Cladribine Tablets: Switch From Oral | Cladribine Tablets: Switch From Infusion
Number analyzed (Participants) | 103 | 85
Participants
  Adverse Event | 9 | 1
  Lost to follow-up | 12 | 6
  Protocol deviation | 4 | 2
  Progressive disease | 1 | 3
  Withdrew consent from study | 9 | 5
  Other/ Not Mentioned | 8 | 2

19. Secondary Outcome: Elapsed Time to Discontinuation After First Dose of Cladribine Tablets
Description: Elapsed time to discontinuation after first dose of cladribine tablets was reported. Elapsed time to discontinuation of cladribine tablets is calculated by subtracting the date of the first study dose from the date on which the participant discontinued cladribine tablets.
Time Frame: Baseline (Month 0) up to 24 Months
Population: The FAS included all participants enrolled in the study who received at least 1 dose of cladribine tablets. "Overall number of participants analyzed" refers to those evaluable for the outcome measure.
Measure: Median (Full Range); unit: months
Arm/Group | Cladribine Tablets: Switch From Oral | Cladribine Tablets: Switch From Infusion
Number analyzed (Participants) | 103 | 80
months | 12.8 [0.0 to 17.4] | 13.1 [0.1 to 22.9]

20. Secondary Outcome: Number of Doses Received by Participants as Per United States Prescribing Information
Description: Number of doses received by participants as per United States prescribing information were reported.
Time Frame: Baseline (Month 0) up to 24 Months
Population: The FAS included all participants enrolled in the study who received at least 1 dose of cladribine tablets.
Measure: Median (Full Range); unit: number of doses received
Arm/Group | Cladribine Tablets: Switch From Oral | Cladribine Tablets: Switch From Infusion
Number analyzed (Participants) | 103 | 85
number of doses received | 24.0 [2.0 to 40.0] | 25.0 [5.0 to 40.0]

21. Secondary Outcome: Total Planned Doses Received by Participants as Per United States Prescribing Information
Description: Total planned doses received by participants as per United States Prescribing Information was reported.
Time Frame: Baseline (Month 0) up to 24 Months
Population: The FAS included all participants enrolled in the study who received at least 1 dose of cladribine tablets.
Measure: Median (Full Range); unit: mg/kg
Arm/Group | Cladribine Tablets: Switch From Oral | Cladribine Tablets: Switch From Infusion
Number analyzed (Participants) | 103 | 85
mg/kg | 3.4 [0.9 to 4.0] | 3.5 [0.9 to 3.9]

22. Secondary Outcome: Percentage of Participants With Subsequent Treatment Chosen Following Discontinuation of Cladribine Tablets
Description: Percentage of participants with subsequent treatment chosen following discontinuation of cladribine tablets was reported. The percentages were calculated using the number of participants who discontinued Cladribine tablets as denominator.
Time Frame: Baseline (Month 0) up to 24 Months
Population: The FAS included all participants enrolled in the study who received at least 1 dose of cladribine tablets.
Measure: Number; unit: percentage of participants
Arm/Group | Cladribine Tablets: Switch From Oral | Cladribine Tablets: Switch From Infusion
Number analyzed (Participants) | 43 | 19
percentage of participants | 4.7 | 5.2

23. Secondary Outcome: Number of Participants With At Least One Concomitant Medication
Description: Number of participants with at least one concomitant medication were reported.
Time Frame: Baseline (Month 0) up to 24 Months
Population: The FAS included all participants enrolled in the study who received at least 1 dose of cladribine tablets.
Measure: Count of Participants; unit: Participants
Arm/Group | Cladribine Tablets: Switch From Oral | Cladribine Tablets: Switch From Infusion
Number analyzed (Participants) | 103 | 85
Participants | 98 | 73

24. Secondary Outcome: Annualized Relapse Rate (ARR)
Description: A relapse was defined as an exacerbation of symptoms that occurred over a minimum of 24 hours and was separated from a previous attack by at least 30 days, in the absence of fever or infection. Annualized relapse rate (ARR) during the 24 months prior to baseline, based on retrospectively collected data, was reported. ARR was calculated as the total number of reported relapses in the 24 months after treatment divided by the days on study corresponding to relapse information and multiplied by 365.25.
Time Frame: Up to 24 Months prior Baseline (Month 0)
Population: The FAS included all participants enrolled in the study who received at least 1 dose of cladribine tablets.
Measure: Mean (Standard Deviation); unit: relapses per year
Arm/Group | Cladribine Tablets: Switch From Oral | Cladribine Tablets: Switch From Infusion
Number analyzed (Participants) | 103 | 85
relapses per year | 0.17 (0.313) | 0.14 (0.268)

25. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs), Adverse Drug Reactions (ADRs) and Adverse Events of Special Interest (AESIs)
Description: A serious adverse event (SAE) is an adverse event (AE) that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect or is otherwise considered medically important. An ADR is a response to a medicinal product which is noxious and unintended. An AESI is an AE of scientific and medical concern specific to the Sponsor's product or program, for which ongoing monitoring and rapid communication by the investigator to the Sponsor can be appropriate. Special Situations included AEs related to pregnancy, overdose, off-label use, misuse, medication error, occupational exposure, or lack of therapeutic effectiveness.
Time Frame: Baseline (Month 0) up to 24 months
Population: The FAS included all participants enrolled in the study who received at least 1 dose of cladribine tablets.
Measure: Count of Participants; unit: Participants
Arm/Group | Cladribine Tablets: Switch From Oral | Cladribine Tablets: Switch From Infusion
Number analyzed (Participants) | 103 | 85
Participants
  TEAEs | 65 | 51
  SAEs | 10 | 14
  ADR | 35 | 19
  AESIs | 15 | 7
  Special Situation | 0 | 4

26. Primary Outcome: Annualized Relapse Rate (ARR)
Description: A relapse was defined as per routine clinical practice as determined by the investigator. As a guide, relapse may be defined as exacerbation of symptoms that occur over a minimum of 24 hours and separated from a previous attack by at least 30 days, in the absence of fever or infection. ARR was calculated as the total number of reported relapses in the 24 months after treatment divided by the days on study corresponding to relapse information and multiplied by 365.25.
Time Frame: From first dose of cladribine tablets up to 24 months
Population: The FAS included all participants enrolled in the study who received at least 1 dose of cladribine tablets.
Measure: Mean (Standard Deviation); unit: relapses per year
Arm/Group | Cladribine Tablets: Switch From Oral | Cladribine Tablets: Switch From Infusion
Number analyzed (Participants) | 103 | 85
relapses per year | 0.04 (0.145) | 0.03 (0.153)

ADVERSE EVENTS:
Time Frame: Baseline (Month 0) up to 24 months
Arm/Group | Cladribine Tablets: Switch From Oral | Cladribine Tablets: Switch From Infusion
All-Cause Mortality (participants affected / at risk) | 2/103 | 0/85
Serious Adverse Events (participants affected / at risk) | 10/103 | 14/85
Other Adverse Events (participants affected / at risk) | 65/103 | 51/85
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cladribine Tablets: Switch From Oral (N=103) | Cladribine Tablets: Switch From Infusion (N=85)
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Breast cellulitis (Infections and infestations) | 1 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 1
COVID-19 (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 2
Sepsis (Infections and infestations) | 0 | 1
Tubo-ovarian abscess (Infections and infestations) | 0 | 1
Ureteritis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Urosepsis (Infections and infestations) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 1
Lymphocyte count decreased (Investigations) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Embolic stroke (Nervous system disorders) | 0 | 1
Optic neuritis (Nervous system disorders) | 0 | 1
Psychogenic seizure (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 0 | 1
Trigeminal neuralgia (Nervous system disorders) | 0 | 1
Abortion threatened (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Drug abuse (Psychiatric disorders) | 0 | 1
Suicide attempt (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Ureterolithiasis (Renal and urinary disorders) | 0 | 2
Urinary tract obstruction (Renal and urinary disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cladribine Tablets: Switch From Oral (N=103) | Cladribine Tablets: Switch From Infusion (N=85)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 20 | 4
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Left ventricular dysfunction (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0
Type V hyperlipidaemia (Congenital, familial and genetic disorders) | 1 | 0
Deafness (Ear and labyrinth disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0
Autoimmune thyroiditis (Endocrine disorders) | 1 | 0
Goitre (Endocrine disorders) | 0 | 1
Hypothyroidism (Endocrine disorders) | 2 | 0
Blindness unilateral (Eye disorders) | 0 | 1
Cataract (Eye disorders) | 1 | 0
Eye pain (Eye disorders) | 1 | 1
Visual impairment (Eye disorders) | 0 | 2
Vitreous opacities (Eye disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1
Anal incontinence (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Dental caries (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 5 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1
Food poisoning (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 2
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Hypoaesthesia oral (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 6 | 2
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1
Adverse drug reaction (General disorders) | 1 | 0
Asthenia (General disorders) | 0 | 1
Fatigue (General disorders) | 9 | 11
Gait disturbance (General disorders) | 0 | 1
Pain (General disorders) | 3 | 0
Peripheral swelling (General disorders) | 1 | 0
Hepatic steatosis (Hepatobiliary disorders) | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1
Conjunctivitis (Infections and infestations) | 0 | 2
Coronavirus infection (Infections and infestations) | 1 | 0
Cystitis (Infections and infestations) | 0 | 1
External ear cellulitis (Infections and infestations) | 0 | 1
Fungal skin infection (Infections and infestations) | 0 | 1
Helicobacter infection (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 1
Nasopharyngitis (Infections and infestations) | 1 | 1
Oral fungal infection (Infections and infestations) | 0 | 1
Oral herpes (Infections and infestations) | 1 | 1
Pneumonia (Infections and infestations) | 1 | 1
Respiratory syncytial virus infection (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 1 | 3
Skin candida (Infections and infestations) | 0 | 1
Subcutaneous abscess (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 4 | 4
Urinary tract infection (Infections and infestations) | 3 | 7
Urinary tract infection fungal (Infections and infestations) | 0 | 1
Vulvovaginal mycotic infection (Infections and infestations) | 1 | 3
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 2
Contusion (Injury, poisoning and procedural complications) | 1 | 2
Fall (Injury, poisoning and procedural complications) | 2 | 4
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1
Joint injury (Injury, poisoning and procedural complications) | 1 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 1
Blood cholesterol increased (Investigations) | 1 | 0
Blood pressure increased (Investigations) | 1 | 0
Liver function test abnormal (Investigations) | 1 | 0
Lymphocyte count decreased (Investigations) | 2 | 1
SARS-CoV-2 test positive (Investigations) | 0 | 1
Weight increased (Investigations) | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Dyslipidaemia (Metabolism and nutrition disorders) | 1 | 0
Glucose tolerance impaired (Metabolism and nutrition disorders) | 1 | 0
Gout (Metabolism and nutrition disorders) | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 1 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 4
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint lock (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 3
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 1
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Altered state of consciousness (Nervous system disorders) | 0 | 1
Amnesia (Nervous system disorders) | 1 | 1
Balance disorder (Nervous system disorders) | 1 | 1
Burning sensation (Nervous system disorders) | 0 | 2
Carpal tunnel syndrome (Nervous system disorders) | 2 | 0
Cognitive disorder (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 2
Facial spasm (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 5 | 3
Hemiparesis (Nervous system disorders) | 0 | 1
Hypoaesthesia (Nervous system disorders) | 4 | 1
Multiple sclerosis relapse (Nervous system disorders) | 2 | 1
Neuralgia (Nervous system disorders) | 0 | 1
Optic neuritis (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 1
Post herpetic neuralgia (Nervous system disorders) | 0 | 1
Radial nerve palsy (Nervous system disorders) | 1 | 0
Restless legs syndrome (Nervous system disorders) | 1 | 0
Sciatica (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 1 | 0
Sensory disturbance (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 0 | 2
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Abnormal dreams (Psychiatric disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 2 | 1
Insomnia (Psychiatric disorders) | 3 | 1
Bladder hypertrophy (Renal and urinary disorders) | 1 | 0
Incontinence (Renal and urinary disorders) | 1 | 0
Micturition urgency (Renal and urinary disorders) | 4 | 0
Pollakiuria (Renal and urinary disorders) | 2 | 1
Ureterolithiasis (Renal and urinary disorders) | 0 | 1
Urethral polyp (Renal and urinary disorders) | 1 | 0
Urinary hesitation (Renal and urinary disorders) | 1 | 0
Breast cyst (Reproductive system and breast disorders) | 1 | 0
Breast pain (Reproductive system and breast disorders) | 1 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 1
Nipple pain (Reproductive system and breast disorders) | 1 | 0
Penile discharge (Reproductive system and breast disorders) | 0 | 1
Perineal pain (Reproductive system and breast disorders) | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 2
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 1
Livedo reticularis (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 1
Aortic dilatation (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1
Essential hypertension (Vascular disorders) | 1 | 0
Hot flush (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 2 | 0
Lymphoedema (Vascular disorders) | 0 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 1
Peripheral coldness (Vascular disorders) | 0 | 1
Peripheral venous disease (Vascular disorders) | 1 | 0
COVID-19 (Infections and infestations) | 8 | 9
Pyelonephritis (Infections and infestations) | 0 | 1
Subclavian artery stenosis (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2024-10-21): https://cdn.clinicaltrials.gov/large-docs/02/NCT03933202/Prot_000.pdf
  • Statistical Analysis Plan (2025-01-23): https://cdn.clinicaltrials.gov/large-docs/02/NCT03933202/SAP_001.pdf